CLINICAL TRIAL: NCT05769764
Title: HER3 Prevalence in Archival Tissue and Associated Real World (RW) Data From Non-Small Cell Lung Cancer Patients
Brief Title: A Study of Prevalence of HER3 Expression in Non-Small Cell Lung Cancer
Status: Completed | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: U31402-0003-NIS-MA
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; HER3 Expression Prevalence; Archival Tissue Samples; Real-World Data
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Archived tissue samples (sourced from biopsies and resections performed as part of routine care) will be procured from Guardian Research Network (GRN) sites for patients who fulfill the study eligibility criteria. These tissue samples will be shipped to a CLIA-certified lab for analysis. De-identified HER3 expression data resulting from testing will be combined with existing clinical data from GRN's electronic medical record (EMR) database.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cohort 1: NSCLC: Participants with NSCLC will be included in this cohort if they do not meet requirements for inclusion in Cohorts 2-4.
  Interventions: Other: Archival tissue specimen and immunohistochemistry staining
- Cohort 2: EGFR-mutated (EGFRm) NSCLC Previously Treated With a 3rd Generation EGFR TKI: Participants with EGFR-mutated (EGFRm) NSCLC previously treated with a 3rd generation tyrosine kinase inhibitor (TKI) with matched samples.
  Interventions: Other: Archival tissue specimen and immunohistochemistry staining
- Cohort 3: ALK+ NSCLC: Participants with ALK+ NSCLC with matched samples.
  Interventions: Other: Archival tissue specimen and immunohistochemistry staining
- Cohort 4: NSCLC Harboring a KRAS p.G12C Mutation or EGFR Exon 20 Insertion: Participants with NSCLC harboring a Kirsten rat sarcoma viral oncogene homolog (KRAS) p.G12C mutation or EGFR exon 20 insertion.
  Interventions: Other: Archival tissue specimen and immunohistochemistry staining

INTERVENTIONS:
Other: Archival tissue specimen and immunohistochemistry staining — This is a non-interventional study and no intervention will be administered.

SUMMARY:
There is currently a lack of published HER3 expression prevalence data among non-small cell lung cancer (NSCLC) patients. The estimation of HER3 expression prevalence in this population using archival tissue samples and the assessment of associated patient characteristics in real world (RW) data will ultimately inform clinical strategy and increase awareness among health care providers (HCPs) and the greater medical community to improve patient care.

DETAILED DESCRIPTION:
The purpose of this study is to use archival tissue samples and RW data to generate HER3 expression prevalence data within the NSCLC population and by patient characteristics (e.g., ethnicity, histology, smoking status, age, prior treatment, etc.).

The primary objective of the study will analyze and assess archival tissue specimens and associated RW data to:

* Increase the understanding of HER3 expression in NSCLC among HCPs and the medical community
* Generate evidence to support future clinical strategies in this area

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years in US
* Histologically or cytologically documented advanced or metastatic NSCLC
* At least one sample available and evaluable for HER3 expression

Additional population-specific inclusion criteria:

For Cohort 1:

* Tissue sample collected on or after January 1, 2013

For Cohort 2:

* EGFRm NSCLC previously treated with a 3rd generation EGFR TKI
* 2 samples are available and evaluable for HER3 expression at 2 timepoints: one pre-treatment and one post-treatment, where the treatment is a 3rd generation TKI (defined as Osimertinib, Aumolertinib [formerly Almonertinib])

For Cohort 3:

* ALK+ NSCLC
* 2 samples are available and evaluable for HER3 expression at 2 timepoints: one pre-treatment and one post-treatment, where the treatment is a TKI

For Cohort 4:

* NSCLC harboring a KRAS p.G12C mutation or EGFR exon 20 insertion
* 2 samples are available and evaluable for HER3 expression at 2 timepoints: one pre-treatment and one post-treatment

Exclusion Criteria:

* Prior treatment with an anti-HER3 antibody or topoisomerase I inhibitor (single-agent or combination)
* Prior treatment with an antibody drug conjugate (ADC) that contains a topoisomerase I inhibitor
* Previous histologic or cytologic evidence of small cell or combined small cell/non-small cell disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The EMR database provided by GRN, an oncology-focused, mission-driven hospital consortium comprised of 37 cancer centers, 85 hospitals and more than two million oncology patients across 13 USA states (New York, Massachusetts, Rhode Island, Maryland, Virginia, South Carolina, Florida, Indiana, Kentucky, Missouri, Arkansas, Kansas, Oklahoma), will be used as the data source for this study.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2022-12-19 (Actual); Primary Completion 2023-04-06 (Actual); Study Completion 2023-04-06 (Actual)

PRIMARY OUTCOMES:
HER3 Expression Prevalence Estimate for the NSCLC Population, Overall | 6 months
  The overall HER3 expression prevalence estimate will be reported.
HER3 Expression Prevalence Estimate for the NSCLC Population, by Subgroup | 6 months
  HER3 expression prevalence estimate will be reported by subgroup, including age, gender, smoking status, epidermal growth factor receptor (EGFR) status, AGA status, ethnicity, and location of biopsy.
HER3 Expression Prevalence Estimate for the NSCLC Population Before and After Treatment, by Patient Subpopulation | 6 months
  HER3 expression prevalence estimate before and after treatment will be reported by patient subpopulation (EGFRm NSCLC previously treated with a 3rd generation EGFR TKI, ALK+ NSCLC, NSCLC harboring a KRAS p.G12C mutation or EGFR exon 20 insertion).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Leader, Study Director — Daiichi Sankyo
Locations (2):
- United States (2):
  - Baptist Health South Florida - Miami Cancer Institute, Miami, Florida
  - McLeod Health, Florence, South Carolina

IPD SHARING:
Plan to Share IPD: No